CLINICAL TRIAL: NCT02875015
Title: Liposomal Bupivacaine vs. Bupivacaine Hydrochloride and Lidocaine During Suburethral Sling Placement: a Randomized Control Trial
Brief Title: Liposomal Bupivacaine vs. Bupivacaine Hydrochloride and Lidocaine During Suburethral Sling Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, charbel salamon, Fellowship Director, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 883788-1
Record Dates: First submitted 2016-06-27; First posted 2016-08-23 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Pain
Keywords: Anesthetics; Anesthetic Effects; Mid-urethral sling
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Lidocaine; Suburethral Slings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal Bupivacaine (Experimental): 20mL of Liposomal Bupivacaine (EXPAREL) will be diluted in 80 mL of injectable saline used for hydro-dissection of the vesicovaginal space and along the track of the sling trocars during the placement of a suburethral sling.
  Interventions: Drug: Liposomal Bupivacaine; Procedure: Suburethral Sling
- Bupivacaine Hydrochloride and Lidocaine (Active Comparator): Bupivacaine Hydrochloride (HCL) and Lidocaine. Fifty mL of 0.05% Marcaine and 30 mL of Lidocaine will be diluted in 100 mL of injectable saline used for hydro-dissection of the vesicovaginal space and along the track of the sling trocars during the placement of a suburethral sling.
  Interventions: Drug: Bupivacaine Hydrochloride and Lidocaine; Procedure: Suburethral Sling

INTERVENTIONS:
Drug: Liposomal Bupivacaine — 20 mL of Liposomal Bupivacaine (EXPAREL) will be diluted in 80 mL of injectable saline used for hydro-dissection of the vesicovaginal space and along the track of the sling trocars
  Other Names: EXPAREL
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine Hydrochloride and Lidocaine — Bupivacaine Hydrochloride (HCL) and Lidocaine. Fifty mL of 0.05% Marcaine and 30 mL of Lidocaine will be diluted in 100 mL of injectable saline used for hydro-dissection of the vesicovaginal space and along the track of the sling trocars during the placement of a suburethral sling.
  Other Names: Marcaine and Lidocaine
  Arms: Bupivacaine Hydrochloride and Lidocaine
Procedure: Suburethral Sling — A retropubic, transobturator or mini-sling will be placed in the usual fashion followed by diagnostic cystoscopy.
  Other Names: Midurethral Sling

SUMMARY:
Postoperative pain, the quality of their recovery and the opioid consumption following a midurethral sling placement are being compared between 2 groups. One group will have the hydro-dissection performed with a diluted liposomal bupivacaine solution. The other group will have the hydro-dissection performed with a diluted bupivacaine HCL and Lidocaine solution.

DETAILED DESCRIPTION:
This is a prospective, comparative, randomized study. Women with pure stress urinary incontinence or mixed urinary incontinence with a predominant stress component who had chosen to proceed with a midurethral sling will be randomized to two groups. The study group will have the hydro-dissection performed with a diluted liposomal bupivacaine solution. The comparison group would have the hydro-dissection performed with a diluted bupivacaine HCL and Lidocaine solution. The postoperative pain will be compared between groups using a visual analog scale. The quality of recovery will be compared between the groups using the quality of recovery short form. Postoperative opioid consumption will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* Age >18 years
* Not Pregnant
* Able to give informed consent
* Electively chose surgical management of SUI with a suburethral sling

Exclusion Criteria:

* Pregnant or nursing
* Allergy to amide anesthetics
* History of drug or alcohol abuse
* Severe cardiovascular, hepatic, renal disease or neurological impairment,
* Long-acting opioid within 3 days or any opioid use within 24 hours before surgery
* Patients taking monoamineoxidase inhibitors (MAOI) or antidepressants of the triptyline or imipramine types
* Contraindication to: Acetaminophen, Non-steroidal anti-inflammatory drugs (NSAID), Hydrocodone, Oxycodone, Hydromorphone AND Morphine,
* Administration of an investigational drug within 30 days before this study
* Chronic pain syndromes
* Daily NSAID or opioid use
* Patients undergoing concomitant procedures

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Postoperative Day 1 Pain | Patient will record her average pain on postop day 1. She will return this result at her postop visit 4-6 weeks after her surgery. These results will be examined and compared at the completion of the study.
  Average pain rating experienced on postoperative day one using the visual analog scale (VAS) on scale of 0 to 10 cm. This will be recorded by the patient prior to going to bed.

SECONDARY OUTCOMES:
Second Stage PACU Postoperative Pain | The PACU nurse will record the patient's pain level upon admission to second stage PACU. These results will be examined and compared at the completion of the study.
  Visual analog scale (VAS) on scale of 0 to 10 cm will be used to evaluate the pain score experienced upon admission to second stage PACU.
Postoperative Pain Upon Discharge | The PACU nurse will record the patient's pain level upon discharge to home. These results will be examined and compared at the completion of the study.
  Visual analog scale (VAS) on scale of 0 to 10 cm will be used to evaluate the pain score experienced upon discharge from the hospital.
Postoperative Pain Four Hours After Discharge | Record the average pain 4 hours after discharge to home. She will return this result at her postop visit 4-6 weeks after her surgery. These results will be examined and compared at the completion of the study.
  Visual analog scale (VAS) on scale of 0 to 10 cm will be used to evaluate the pain score experienced. This will be recorded 4 hours after being discharged from the hospital.
Night of Surgery Postoperative Pain | Pt will record her average pain on the night of surgery. She will return this result at her postop visit which is approximately 4-6 weeks after her surgery. These results will be examined and compared at the completion of the study.
  Visual analog scale (VAS) on scale of 0 to 10 cm will be used to evaluate the pain score experienced that day and recorded prior to going to bed on the night of surgery.
Postoperative Days 2 through 7 Pain | Pt will record her average pain from postop days 2-7. She will return this result at her postop visit 4-6 weeks after her surgery. These results will be examined and compared at the completion of the study.
  Visual analog scale (VAS) on scale of 0 to 10 cm will be used to evaluate the pain score experienced that day and recorded prior to going to bed on postop days 2-7.
Preoperative Quality of Recovery | The patient will complete the questionnaire prior to surgery. This will be collected prior to surgery. These results will be examined and compared at the completion of the study.
  Baseline Quality of Life and Recovery as measured by the ambulatory QoR15 preoperatively on the day of surgery.
Postoperative Days 1, 7 and 14 Quality of Recovery | The patient will complete the questionnaire on postop days 1, 7 & 14. She will return these results at her postop visit 4-6 weeks after her surgery. These results will be examined and compared at the completion of the study.
  Quality of Life and Recovery as measured by the ambulatory QoR15 on postoperative days 1, 7 and 14.
Postoperative Narcotic Consumption | The patient will record narcotic consumption each day from the day of surgery to postop day 7. She will return this result at her postop visit 4-6 weeks after her surgery. These results will be examined and compared at the completion of the study.
  The total amount of narcotic taken the night of surgery and each day thereafter through postoperative day seven will be recorded each night prior to going to bed.

CONTACTS AND LOCATIONS:
Overall Officials: Charbel Salamon, MD, Principal Investigator — Atlantic Health System
Locations (2):
- United States (2):
  - Morrristown Medical Center, Morristown, New Jersey
  - Overlool Medical Center, Summit, New Jersey

IPD SHARING:
Plan to Share IPD: No